CLINICAL TRIAL: NCT02211547
Title: Effect of Low Level Laser Therapy on Pain Induced by Placement of Orthodontic Separators in Pediatric Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 13-3091
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Levels of Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): No treatment to be rendered following separator placement.
- Placebo (Placebo Comparator): Single blind lack of laser treatment (the laser will be positioned and operated as if applying the treatment, but the energy transfer will not take place).
  Interventions: Other: Placebo
- Treatment (Experimental): Single blind laser treatment (the laser will be positioned and operated, and energy transfer will take place).
  Interventions: Device: Epic 10 Diode Laser by Biolase Inc.

INTERVENTIONS:
Device: Epic 10 Diode Laser by Biolase Inc.
  Other Names: Epic 10 Diode Laser by Biolase Inc. (Irvine, CA); Product Code: GEX,ILY; Regulatory Class: II; Regulation number: 878.4810, 510(K); Number: K121286, with an InGaAsP diode, frequency of 50 Hz, wavelength of 940 nm, and output potency of 10 watts.
  Arms: Treatment
Other: Placebo — Single blind lack of laser treatment (the laser will be positioned and operated as if applying the treatment, but the energy transfer will not take place).
  Arms: Placebo

SUMMARY:
The primary goal of the study is to determine if there is a difference in pain levels following the use of low level laser therapy versus placebo and control after placement of elastomeric orthodontic separators in pediatric patients. To test this, the investigators will assess the patient's pain levels immediately following separator placement and 24 hours post-operatively but having patients rate their pain on a 10 cm Visual Analog Scale (VAS). Patients will be randomly assigned to one of three groups: treatment, placebo, and control. The aim of this study is to establish whether or not low level laser therapy can be used to reduce pain in pediatric patients following separator placement.

ELIGIBILITY:
Inclusion Criteria:

* Absence of acute or chronic dental disease and periodontal disease
* Free from severe systemic disease
* No fixed orthodontic appliances currently placed
* No ankylosis or tooth implants within dentition
* No analgesic drug consumption for 48 hours preceding the study and during the study, a minimum age of 6 years

Exclusion Criteria:

* Presence of a diastema where the separator would be placed
* Conditions that could alter nociception, such as current or previous use of anti-inflammatory and analgesic drugs, antidepressants, anticonvulsants, and oral contraceptives
* Any medical conditions or medications that may contraindicate use of certain light/laser sources such as low level laser therapy (LLLT)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Pain experienced by the patient | 24 hours
  Pain will be assessed via a 10 cm non-hashed visual analog scale at two time points, immediately after placement of the elastomeric separators (time 0), and approximately 24 hours after placement when the patient returns to the clinic for separator removal.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Murzyn-Dantzer, DMD,MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Pediatric Dental Center, Aurora, Colorado, United States